CLINICAL TRIAL: NCT03034304
Title: Multi-center, Phase I Clinical Study to Evaluate the Safety and Tolerability of Multiple Antigen Stimulating Cellular Therapy-I (MASCT-I) in Patients With Advanced Solid Tumor, and to Preliminarily Evaluate the Anti-tumor Efficacy of MASCT-I Alone, in Combination With Chemical Drugs, and in Combination With PD1 Antibody
Brief Title: A Phase I Clinical Study for Evaluating the Safety and Efficacy of MASCT-I in Patients With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated early due to the COVID-19 pandemic and sponsor's funding constraints, based on promising preliminary safety and efficacy data.
Sponsor: HRYZ Biotech Co. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRYZ MASCT-I-1001
Record Dates: First submitted 2016-12-26; First posted 2017-01-27 (Estimated); Last update posted 2025-07-24 (Actual); Status verified 2025-05

CONDITIONS: Advanced Solid Tumors
Keywords: MASCT-I,DC,T cell; Advanced solid tumors
MeSH Terms: interventions — Ifosfamide; spartalizumab; Doxorubicin; Gemcitabine; Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MASCT-I alone or in combination with chemical drugs or in combination with PD-1 antibody (Experimental): Group 1: MASCT-I alone;
  Group 2: Advanced urothelial carcinoma and cholangiocarcinoma treatment with MASCT-I alone,Advanced soft tissue sarcoma and osteosarcoma treatment with MASCT-I alone or combination with ifosfamide. In the event of disease progression, treatment with MASCT-I +PD1 antibody;
  Group 3: Advanced metastatic or recurrent urothelial carcinoma, soft tissue sarcoma/osteosarcoma, and cholangiocarcinoma that progressed after first line chemotherapy were treated with MASCT-I combined with PD1 antibody;
  Group 4: Recurrent metastatic solid tumors that had failed previous treatment with PD1 antibody were treated with MASCT-I + PD1 antibody;
  Group 5: Untreated advanced soft tissue sarcom treatment with MASCT-I+AI (Adriamycin+ifosfamide);
  Group 6: Untreated advanced urothelial carcinoma treatment with MASCT-I+GP/GC(Gemcitabine+cisplatin/ Gemcitabine+carboplatin);
  Interventions: Biological: MASCT-I; Drug: Ifosfamide; Drug: PD1 antibody; Drug: Adriamycin; Drug: Gemcitabine; Drug: Cisplatin; Drug: Carboplatin

INTERVENTIONS:
Biological: MASCT-I — The final products of MASCT-I technology are dendritic cells (DC) and effector T cells
Drug: Ifosfamide — 2g/m2/d, intravenous drip for 30min. Administration is conducted for continuous 5 days. After 4 weeks, the above cycle is repeated for 6 continuous cycles
Drug: PD1 antibody — 200 mg/every two weeks ,four weeks is a cycle. Subjects were treated with MASCT-I combined with PD1 antibody until disease progression, MASCT-I intolerance or study completion. If PD1 antibody intolerance occurs, MASCT-I therapy alone will continue. MASCT-I and PD1 antibody are adminnistered according to their respective drug cycle without interfering with each other.
Drug: Adriamycin — 60mg/m2, from the first day of each cycle, it is used for 1-2 days, intravenous drip. Repeat the above cycle after 4 weeks, no more than 8 cycles
Drug: Gemcitabine — 1000 mg/m2, Intravenous drip for about 30 min, used on the first and eighth days of each cycle, and every 3-4 weeks as a cycle
Drug: Cisplatin — 70mg/m2, Use on the first day of each chemotherapy cycle, intravenous drip for 30-120 min, and every 3-4 weeks as a cycle;
Drug: Carboplatin — 5mg/ml/min, Use it on the first day of each chemotherapy cycle, intravenous drip for 30 minutes, and every 3-4 weeks as a cycle

SUMMARY:
The purpose of this study is to evaluate Safety and tolerability of MASCT-I in patients with advanced solid tumors, either alone or in combination with chemical drugs or in combination with PD1 antibody.

DETAILED DESCRIPTION:
The multiple-antigen specific cell therapy which was developed by Hengrui Yuanzheng is optimized continuously and has been upgraded from the first-generation MASCT technology to MASCT-I. MASCT-I is a technology which add PD1 antibody in vitro cell culture process of MASCT cell culture to block PD1 receptor on immunocytes, release the brake on immunocytes' reinfusion and interaction with tumor cells for enhancing the efficacy of immunocytes' killing tumor cells. At present, the development and validation of manufacturing process has been completed, and it is urgently needed to conduct the validation of clinical effect.

This is a Multi-center, phase I clinical study to evaluate the safety and tolerability of multiple antigen stimulating cellular therapy-I (MASCT-I) in patients with advanced solid tumor, and to preliminarily evaluate the anti-tumor efficacy of MASCT-I alone, in combination with chemical drugs, and in combination with PD1 antibody. About 193 cases of adult patients with advanced solid tumors will be recruited.

ELIGIBILITY:
Major Inclusion Criteria:

1. Age 18-70 at screening;
2. Obtain written informed consent of the subject/legal representative prior to conducting any program related procedures, including evaluation during the screening period;
3. Scored 0 -1 on ECOG;
4. Life expectancy ≥6 months;
5. Cardiopulmonary function is basically normal;
6. Results of blood test and biochemistry at baseline meeting the following criteria:Hemoglobin≥85g/L,Leucocyte≥3.0×109/L,Absolute neutrophil count(ANC)≥1.5×109/L,Trombocyte≥70×109/L,ALT/AST ≤ 2.5×ULN or ≤ 5×ULN for patients with hepatic metastases, ALP≤2.5 times of upper limit of normal, Serum total bilirubin < 1.5×ULN,Serum urea nitrogen and creatinine ≤ 1.5×ULN,patients with urothelial carcinoma,Serum urea nitrogen and creatinine ≤ 2.5×ULN, Serum albumin ≥30g/L

For the first group of subjects, the following criteria should be met:

1. Patients who suffer from advanced (unresectable) or recurrent solid tumors (only limited to bladder cancer and soft tissue sarcoma) confirmed by histology and cytology and are treated unsuccessfully with various standard therapies;
2. According to RECIST1.1 criteria, there must be one measurable focus;
3. Time interval between end of other anti-tumor measures and this study treatment is at least 1 month;

For the second group of subjects, the following criteria should be met:

1. Urothelial carcinoma: histologically or cytologically confirmed that gemcitabine + platinum-based first-line chemotherapy achieved clinical benefit after 4-6 cycles of advanced recurrence or metastasis;
2. Soft tissue sarcoma or osteosarcoma: Subjects who histologically or cytologically demonstrated clinical benefit after at least 4 cycles of doxorubicin-based first-line chemotherapy following advanced recurrence or metastasis. For some subjects who are intolerant or insensitive to chemotherapy, screening can also be conducted after other first-line treatment regiments achieve clinical benefit.
3. Cholangiocarcinoma: Histologically or cytologically confirmed, first-line treatment after advanced recurrence or metastasis is beneficial.

Note: Clinical benefit is defined as complete response (CR), partial response (PR), or disease stabilization (SD). The disease stabilizes for more than 2 months.

For subjects in the third group, the following criteria should be met:

1. Urothelial carcinoma: histologically or cytologically confirmed disease progression after advanced recurrence or metastasis following gemcitabine + platinum regimen first-line chemotherapy;
2. Soft tissue sarcoma or osteosarcoma: histologically or cytologically confirmed disease progression after advanced recurrence or metastasis followed by first-line chemotherapy dominated by adriamycin; For some subjects who are intolerant or insensitive to chemotherapy, they can also be screened after other first-line treatment regiments fail.
3. Cholangiocarcinoma: histologically or cytologically confirmed, progression after first-line treatment after advanced recurrence or metastasis;
4. According to RECIST1.1, at least one measurable lesion must be present;
5. An interval of at least 4 weeks between the end of other anticancer treatments and the treatment in this study;

For the fourth group of subjects, the following criteria should be met:

1. Solid tumor with advanced recurrence or metastasis;
2. PD1 antibody therapy has been used before, and the disease is progressing. The interval between the end of PD1 antibody therapy and this study is at least 4 weeks;
3. According to RECIST1.1, at least one measurable lesion must be present;
4. The interval between the end of other anticancer treatments and the treatment in this study should be at least 4 weeks;

For the fifth group of subjects, the following criteria should be met:

1. Subjects with pathologically confirmed soft tissue sarcoma, locally advanced or metastatic, and inoperable, have not undergone systemic treatment;
2. According to RECIST1.1, at least one measurable lesion must be present

For the sixth group of subjects, the following criteria should be met:

1. Histologically or cytologically confirmed inoperable locally advanced or metastatic urothelial carcinoma (T4b, any N; Or any T, N 2-3) or metastatic urothelial carcinoma (M1, stage IV) including renal pelvis, ureter, bladder, and urethra);
2. Had not previously received systemic chemotherapy for locally advanced or metastatic urothelial carcinoma (UC);
3. At least one measurable lesion was evaluated (based on RECIST1.1 criteria); If the measurable lesion has previously undergone radiotherapy, it needs to be clearly documented that it is now a lesion after disease progression.
4. For subjects who had previously received local intravesical infusion chemotherapy or immunotherapy, this local therapy needed to be completed at least 4 weeks prior to the initiation of the first chemotherapy in this trial
5. Glomerular filtration rate ≥30ml/ min (creatinine clearance was calculated using the standard Cockcroft-Gault formula);

Major Exclusion Criteria:

1. Subjects have clinically manifested central nervous system metastases (such as brain edema, need for hormonal intervention, or progression of brain metastases). Subjects who have received previous treatment for brain or meningeal metastasis, such as clinical stability (MRI) for at least 2 months, and have ceased systemic sex hormone therapy (>10mg/ day prednisone or other therapeutic hormones) for more than 2 weeks may be included;
2. Subjects are receiving immunosuppressive, or systemic, or absorbable local hormone therapy for immunosuppression purposes (>10mg/ day prednisone or other therapeutic hormones) and continue to receive such therapy within 2 weeks prior to enrollment;
3. Subjects are taking immunomodulator drugs and continue to use them within 2 weeks prior to enrollment;
4. Subjects have received MASCT or other cellular immunotherapy or PD1 antibody therapy in the previous year (subjects in the fourth group are not limited to PD1 antibody therapy);
5. Subject has any active autoimmune disease or a history of autoimmune disease;
6. The subject has active tuberculosis;
7. Subject has hepatitis C or HIV infection, or syphilis infection;
8. Patients with gastrointestinal stromal tumor, Ewing sarcoma and rhabdomyosarcoma
9. Patients with recurrence or metastasis during the adjuvant treatment after radical surgery or within 6 months after the end of the treatment (only for patients in Group 5 and Group 6):
10. Those who have used targeted therapy, radiotherapy, immunotherapy or other treatment schemes with clear anti-tumor effect within 4 weeks before enrollment, such as arrotinib, gemcitabine and traditional Chinese medicine; However, if the focus of radiotherapy is not a target focus or there is clear progress after radiotherapy, it can be considered to be included in the group (only for the fifth and sixth groups of subjects);
11. Those who are not suitable for treatment with A1 scheme (only for the fifth group of subjects)
12. Hearing impairment with CTCAE grade>2 (for the sixth group)
13. Peripheral neuropathy with CTCAE grade >2 (such as sensory degeneration, sensory abnormality, including tingling sensation) (for the sixth group);
14. The investigators believed that the subjects were not suitable for chemotherapy containing platinum or gemcitabine (for the sixth group);

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2017-02-22 (Actual); Primary Completion 2023-11-13 (Actual); Study Completion 2023-11-13 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events(Safety) | up to 96 weeks
  All the local reactions, systemic reactions, adverse events and serious adverse events of all the patients will be collected from the informed consent to the end of the study.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events(Safety) | up to 96 weeks
  All the local reactions, systemic reactions, adverse events and serious adverse events of all the patients will be collected from the the informed consent to the end of the study.
Disease Control Rate (DCR) | up to 96 weeks
  Disease control rate is defined as the number of patients with a best overall response of complete response (CR), partial response (PR), or stable disease (SD) based on RESIST v1.1 criteria
Progression-Free Survival (PFS) | up to 96 weeks
  The length of time from enrollment until the time of progression of disease
Overall Survival (OS) | up to 96 weeks
  From enrollment to death of patients
Time to recurrence (TTR) | up to 96 weeks
  the period of time from signing of the ICF by the patient to progression of tumor
time to progression(TTP) | up to 96 weeks
  Time from the first successful apheresis to the first progression of the tumor.
Objective response rate | up to 96 weeks
  The percentage of subjects with PR or CR.

CONTACTS AND LOCATIONS:
Overall Officials: Ruihua Xu, Doctor, Principal Investigator — Sun Yat-sen University
Locations (9):
- China (9):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Zhongshan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality
  - Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality
  - Tianjin Cancer Hospital, Tianjin, Tianjin Municipality
  - The Second Affiliated hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Tumor Hospita, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided